CLINICAL TRIAL: NCT03814811
Title: Circulating Osteocalcin-positive Cells as a Cell-Based Biomarker of Breast Cancer Bone Metastasis Progression
Brief Title: Circulating Osteocalcin-positive Cells in Breast Cancer Bone Metastasis
Acronym: COP-BREAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government)
Responsible Party: Sponsor
Other Study IDs: SNUH-IRB-1706069859
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Breast Neoplasms; Bone Metastases
Keywords: Breast Cancer; Bone; Metastasis; Osteoblast
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Cell Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Bone metastasis(+) with low cOC: Patients who have bone metastasis with low number of circulating osteocalcin-positive (cOC) cells
  Interventions: Diagnostic Test: Circulating Osteocalcin-positive (cOC) cells
- Bone metastasis(+) with high cOC: Patients who have bone metastasis with high number of circulating osteocalcin-positive (cOC) cells
  Interventions: Diagnostic Test: Circulating Osteocalcin-positive (cOC) cells
- Bone metastasis(-) with low cOC: Patients who have metastasis only in extraskeletal sites with low number of circulating osteocalcin-positive (cOC) cells
  Interventions: Diagnostic Test: Circulating Osteocalcin-positive (cOC) cells
- Bone metastasis(-) with high cOC: Patients who have metastasis only in extraskeletal sites with high number of circulating osteocalcin-positive (cOC) cells
  Interventions: Diagnostic Test: Circulating Osteocalcin-positive (cOC) cells

INTERVENTIONS:
Diagnostic Test: Circulating Osteocalcin-positive (cOC) cells — Quantitative measurement of osteocalcin-positive cells in the peripheral blood mononuclear cells by flow cytometry

SUMMARY:
Bone metastasis (i.e. cancer cell spreading to bone) is the major clinical problem of advanced breast cancer patients. Bone metastasis is not curable nor preventable. Currently available therapeutic approaches are only palliative. The major hurdle for improving bone metastasis treatment is lack of sensitive diagnostic tools. Diagnosis of bone metastasis is heavily dependent on radiographic imaging of bone destruction that are detectable only when the lesion is significantly large. Accordingly, if bone metastasis can be detected at an earlier time point when bone destruction is minimal or incipient, treatments can be given earlier and the patients can expect better outcomes. We and others previously have found that a subset of bone-forming cells (i.e. circulating osteocalcin-positive cells) exists in the blood stream of the patients with bone diseases (e.g. bone metastasis and inflammation) or active bone formation (e.g. adolescence) in mouse models anf human samples. Extended from this laboratory observation, this clinical study proposes to test the hypothesis that circulating osteocalcin-positive cells are the early biomarker of breast cancer bone metastasis. For this aim, this study will measure circulating osteocalcin-positive cells in the blood samples of breast cancer patient, and examine whether the measure sensitively detects bone metastasis.

DETAILED DESCRIPTION:
Bone is the most common site of breast cancer metastasis, and the skeletal-related events (SRE) of bone metastasis such as pathologic fractures, cord compression, hypercalcemia and severe pain, accounting for poor quality of life in the terminal stage of the afflicted patients. Since previous SREs are the major risk factors for subsequent SREs related to serious morbidity and mortality, the early detection of bone metastasis prior to clinical symptoms is essential to the better management of breast cancer patients. Currently, diagnosis of bone metastasis is dependent on imaging modalities such as whole-body bone scintigraphy (WBBS). However, detectability of radionuclide activity in the WBBS depends on gross structural bone destruction resulting from considerable progression of macro-metastasis.

Circulating osteoprogenitor cells that is defined a small monocytic cells expressing osteocalcin, a late osteoblast differentiation marker, had been identified in human peripheral blood mononuclear cells (PBMCs). Flow cytometric analyses of the PBMCs using anti-osteocalcin antibody demonstrated that adolescents who are in the period of rapid bone growth showed higher fractions of osteocalcin-positive cells than adults. Moreover, these cells also positively correlated with pathologic changes of bone turnover in such conditions as fracture, hypoparathyroidism, or diabetes. Collectively, circulating osteoprogenitor cells reflects changes of bone turnover in either physiologic or pathologic status.

The scientific hypothesis of this study is that circulating osteoprogenitor cells increases in the early phase of bone micro-metastasis, and the aim of this clinical study is to investigate the difference of circulating osteoprogenitor cells in metastatic breast cancer with or without bone metastasis. This study will also examine whether the patients who have higher number of osteocalcin-positive cells develop bone metastasis at an earlier time point, to validate the value of circulating osteoprogenitor cells in monitoring and/or predictinng the progression of bone metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Stages 2A-4 breast cancer patients who are subject to adjuvant chemotherapy or radiotherapy
* 20 years of age or greater
* Female
* Ability to understand the study objectives and willingness to sign written consent
* ECOG status 0, 1 or 2

Exclusion Criteria:

* History of primary cancer diagnosis in other sites than breast within 5 years
* Diseases of bone metabolism including primary hyperparathyroidism, Paget's disease, osteomalacia, osteogenesis imperfecta
* ECOG status 3 or 4
* Retraction of written consent

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females are eligible.
Study Population: * Patients in Seoul National University Hospital or Korea University Anam Hospital, Seoul, Korea
  * Residents of the Republic of Korea
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression of bone metastasis | 18 months after enrollment
  Metastatic bone lesions will be re-evaluated at 18 months using imaging studies such as bone scan, CT, MRI, or PET or incidence of active skeletal-related events (SREs) such as pathologic fracture or progressive neurologic signs
Diagnosis of new bone metastasis | 18 months after enrollment
  De novo bone metastasis will be diagnosed using imaging studies

CONTACTS AND LOCATIONS:
Overall Officials: Sun Wook Cho, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong HM, Cho SW, Park SI. Osteoblasts Are the Centerpiece of the Metastatic Bone Microenvironment. Endocrinol Metab (Seoul). 2016 Dec;31(4):485-492. doi: 10.3803/EnM.2016.31.4.485. PMID 28029019
- [Background] Eghbali-Fatourechi GZ, Lamsam J, Fraser D, Nagel D, Riggs BL, Khosla S. Circulating osteoblast-lineage cells in humans. N Engl J Med. 2005 May 12;352(19):1959-66. doi: 10.1056/NEJMoa044264. PMID 15888696
- [Background] Gabrilovich DI, Nagaraj S. Myeloid-derived suppressor cells as regulators of the immune system. Nat Rev Immunol. 2009 Mar;9(3):162-74. doi: 10.1038/nri2506. PMID 19197294
- [Background] Manavalan JS, Cremers S, Dempster DW, Zhou H, Dworakowski E, Kode A, Kousteni S, Rubin MR. Circulating osteogenic precursor cells in type 2 diabetes mellitus. J Clin Endocrinol Metab. 2012 Sep;97(9):3240-50. doi: 10.1210/jc.2012-1546. Epub 2012 Jun 27. PMID 22740707